CLINICAL TRIAL: NCT02371642
Title: The Utility of Strain Echocardiography in the Management of Acute Heart Failure
Brief Title: Strain Echo in Acute Heart Failure
Acronym: Strain Echo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Favot, MD, Assistant Professor of Emergency Medicine, Wayne State University
Other Study IDs: unsponsored
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this project is to evaluate the utility of left ventricular strain as part of the assessment of patients in the emergency department with acute heart failure (HF). The central hypothesis of the investigation is that left ventricular strain will prove to be a treatment response variable in patients with acute HF. Patients who are being treated for acute HF with intravenous (IV) vasoactive medications (diuretics, vasodilators, inotropes) will be eligible for enrollment. Patients who give written consent will receive a focused bedside echocardiogram within 30 minutes of the initiation of therapy for acute HF. Images that are captured during this echocardiogram will be interpreted by a blinded cardiologist offline. 23 hours after this initial focused echocardiogram a member of the study team will perform a follow-up focused echocardiogram, capturing the same images that will then be interpreted by a blinded cardiologist offline.

Offline analysis will be performed using a proprietary software package from General Electric called Automated Function Imaging (AFI). The AFI software will be used to calculate longitudinal strain of the left ventricle (LV). Regional and global strain values will be calculated for each focused echocardiogram for each subject. It is our hypothesis that LV strain will demonstrate improvements from the initial echocardiogram to the follow-up echocardiogram, unlike other echocardiographic indices in HF such as LV ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Ability for the patient to provide written informed consent
* Planned treatment with intravenous (IV) medications (diuretics, vasodilators, inotropes) for acute HF

Exclusion Criteria:

* Need for emergent, resuscitative intervention (e.g., cardiopulmonary resuscitation, endotracheal intubation)
* Rapid atrial fibrillation or other arrhythmia that requires IV rate or rhythm control
* Plans for emergent percutaneous coronary intervention (PCI) from the ED
* Pregnancy
* Incarceration
* history of cardiac transplant
* planned transfer to another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be recruited in the emergency department (ED) of Detroit Receiving Hospital (DRH). The DRH ED has research team coverage 24 hours a day, 7 days a week and existing research personnel will be specifically trained to assist with subject identification for this protocol. We will also utilize resident physicians who are on ED based ultrasound and critical care rotations to help identify potential subjects and ensure that participants are captured early in their course and prior to initial treatment for acute HF. The ED will have 2 emergency ultrasound fellows beginning in July 2014 who will also assist with patient recruitment and performance of bedside echocardiograms for purposes of the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
change in global longitudinal strain (GLS) | 23 hours

SECONDARY OUTCOMES:
Readmission rate | 30 days
  Readmission for heart failure or other cardiovascular-related events

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Receiving Hospital, Detroit, Michigan, United States